CLINICAL TRIAL: NCT02851810
Title: Oculomotor and Neurophysiological Markers of Emotion Regulation and Attachment Styles in Adolescence
Brief Title: Oculomotor Markers and Attachment in Adolescents
Acronym: MONRADO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: API/2012/35
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Emotion Dysregulation
Keywords: attachment; oculomotor marker; emotion regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: oculomotor parameter recording — visual scanning behavior is assessed during visualization of emotional pictures
Behavioral: attachment scale interview (ASI) — ASI is used to determine the attachment style of each participant
Behavioral: psychophysiological recording — this consists of the measurement of the skin conductance reactivity (SCR) during the picture visualization
Behavioral: psychometric assessment — self administered questionnaires are used to assess anxiety, depression and alexithymia.
Behavioral: parent interview — an interview of the adolescent parent is performed in order to assess the confusion of the parent-child role and the interaction between the child and its parent.

SUMMARY:
The study aims to identify specific visual scanning patterns of attachment pictures in adolescent with different attachment style.

DETAILED DESCRIPTION:
Oculomotor parameters will be assessed during visualization of 2 sets of pictures. The first set presents a distress picture and is followed by a slide composed of 3 pictures (one representing comfort, one representing complicity and the last representing a neutral scene).

Psychophysiological parameters (skin conductance reactivity-SCR) is also assess during this visualization.

ELIGIBILITY:
Inclusion Criteria:

* non hospitalized child who is going to school

Exclusion Criteria:

* not french-speaker vision problem more than 20 cigarettes/day

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
number of entry in distress pictures | within 1 year after inclusion
  these parameters will be compared between the different types of attachment.
saccade duration in distress picture | within 1 year after inclusion
  time spent looking at the distress picture these parameters will be compared between the different types of attachment.
average of the number of entry in comfort picture vs neutral and complicity pictures | within 1 year after inclusion
  these parameters will be compared between the different types of attachment.
average of the saccade duration in comfort picture vs neutral and complicity pictures | within 1 year after inclusion
  these parameters will be compared between the different types of attachment.

SECONDARY OUTCOMES:
Amplitude of SCR | within 1 year after inclusion
  this parameter will be compared between the different types of attachment.
interaction with the parent: score to the GPACS (goal-corrected partnership in adolescence coding system) | within 1 year after inclusion
  the quality of the interaction with the parent and the confusion of the parent-child role will be compared between the different attachment types.
Reaction time in SCR | within 1 year after inclusion
  this parameter will be compared between the different types of attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane Vulliez-Coady, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szymanska M, Monnin J, Tio G, Vidal C, Girard F, Galdon L, Smith CC, Bifulco A, Nezelof S, Vulliez-Coady L. How do adolescents regulate distress according to attachment style? A combined eye-tracking and neurophysiological approach. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:39-47. doi: 10.1016/j.pnpbp.2018.08.019. Epub 2018 Aug 27. PMID 30165119